CLINICAL TRIAL: NCT00532935
Title: A Phase III Randomized, Active-Comparator (Pioglitazone) Controlled Clinical Trial to Study the Efficacy and Safety of the MK0431A (A Fixed-Dose Combination Tablet of Sitagliptin and Metformin) in Patients With Type 2 Diabetes Mellitus
Brief Title: MK0431A vs. Pioglitazone in Patients With Type 2 Diabetes Mellitus (0431A-066)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431A-066; 2007_510
Record Dates: First submitted 2007-09-19; First posted 2007-09-21 (Estimated); Results first posted 2010-10-18 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination; Pioglitazone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Sitagliptin phosphate (+) metformin hydrochloride
  Interventions: Drug: sitagliptin phosphate (+) metformin hydrochloride
- 2 (Active Comparator): pioglitazone
  Interventions: Drug: Comparator: pioglitazone

INTERVENTIONS:
Drug: sitagliptin phosphate (+) metformin hydrochloride — sitagliptin phosphate (+) metformin hydrochloride 50/500 mg tablet bid, titrating up to sitagliptin phosphate (+) metformin hydrochloride 50/1000 mg tablet for an ~32 wk treatment period
  Other Names: Janumet
  Arms: 1
Drug: Comparator: pioglitazone — pioglitazone 30 mg tablet qd, titrating up to 45 mg qd for an ~32-wk treatment period.
  Other Names: pioglitazone
  Arms: 2

SUMMARY:
A study to evaluate the efficacy and safety of MK0431A in comparison to a commonly used medication in patients with type 2 diabetes

ELIGIBILITY:
General Inclusion Criteria:

* Patient has type 2 diabetes mellitus
* Patient is inadequately controlled and not on treatment with insulin or oral antihyperglycemic therapy

General Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or history of ketoacidosis
* Patient was on antihyperglycemic agent therapy (oral or insulin) within the prior 12 weeks
* Patient was on >4 weeks (cumulatively) of antihyperglycemic therapy (oral or insulin) over the prior 3 years

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2008-01-26 (Actual); Primary Completion 2009-10-23 (Actual); Study Completion 2009-10-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Wainstein J, Katz L, Engel SS, Xu L, Golm GT, Hussain S, O'Neill EA, Kaufman KD, Goldstein BJ. Initial therapy with the fixed-dose combination of sitagliptin and metformin results in greater improvement in glycaemic control compared with pioglitazone monotherapy in patients with type 2 diabetes. Diabetes Obes Metab. 2012 May;14(5):409-18. doi: 10.1111/j.1463-1326.2011.01530.x. Epub 2011 Dec 22. PMID 22059736

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 19-Mar-2008
  Last Patient Last Visit: 23-Oct-2009
  Seventy-four medical clinics worldwide (19 sites in the United States, 31 in Eastern Europe, and 24 in the rest of the world).
Pre-assignment Details: Patients 18-78 years old with Type 2 Diabetes Mellitus (T2DM), drug-naïve (off antihyperglycemic agent
  [AHA] for at least 3 months prior to screening, and a maximum 4 weeks cumulative AHA therapy over the
  previous 3 years), hemoglobin A1C 7.5 to 12% were eligible. Eligible patients underwent a 2-week placebo
  run-in period prior to randomization.
Groups:
- Sitagliptin/Metformin Fixed-Dose Combination: The Sitagliptin/Metformin Fixed-Dose Combination (Sita/Met FDC) group includes data from patients randomized to receive treatment with oral tablets of Sita/Met FDC initiated at a dose of 50/500 mg twice a day (b.i.d). The dose was to have been up-titrated over 4 weeks to 50/1000 mg b.i.d. Patients were discontinued if they were considered clinically inappropriate for up-titration or could not be up-titrated or maintained on the up-titrated dose.
- Pioglitazone: The Pioglitazone group includes data from patients randomized to receive treatment with oral tablets of pioglitazone initiated at a dose of 30 mg once daily (q.d.). The dose was to have been up-titrated over 4 weeks to 45 mg q.d. Patients were discontinued if they were considered clinically inappropriate for up-titration or could not be up-titrated or maintained on the up-titrated dose.
Period: Overall Study
Arm/Group | Sitagliptin/Metformin Fixed-Dose Combination | Pioglitazone
Started | 261 (Excludes 1 patient who was randomized twice at different sites.) | 256 (Excludes 1 patient who was randomized twice at different sites.)
Completed | 210 | 204
Not Completed | 51 | 52
Not completed — Adverse Event | 11 | 12
Not completed — Lack of Efficacy | 0 | 3
Not completed — Lost to Follow-up | 10 | 6
Not completed — Physician Decision | 4 | 5
Not completed — Pregnancy | 1 | 0
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 10 | 9
Not completed — Protocol Specific Criteria | 11 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin/Metformin Fixed-Dose Combination | Pioglitazone | Total
Number analyzed (Participants) | 261 | 256 | 517
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.4 (10.7) | 52.2 (11) | 52.3 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 122 | 240
  Male | 143 | 134 | 277
Race/Ethnicity, Customized [Number; unit: participants]
  White | 168 | 167 | 335
  Black | 6 | 5 | 11
  American Indian | 2 | 0 | 2
  Asian | 58 | 55 | 113
  Multi-racial | 27 | 29 | 56
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent of glycosylated hemoglobin (A1C)] | 9.0 (1.3) | 8.9 (1.3) | 8.9 (1.3)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] | 190.6 (53.4) | 188.9 (57.1) | 189.8 (55.2)
2-Hour Post-Meal Glucose (2-HR PMG) [Mean (Standard Deviation); unit: mg/dL] | 273.7 (84.8) | 278.8 (86.4) | 276.2 (85.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 32
Description: A1C is measured as a percent. Thus this change from baseline reflects the Week 32 A1C percent minus the baseline A1C percent
Time Frame: Baseline and Week 32
Population: The Full Analysis Set (FAS) included all patients who received at least one dose of double-blind study drug and had both a baseline value and ≥ 1 post-baseline value for this outcome. For FAS patients with no data at Week 32, the last non-baseline observed measurement was carried forward to Week 32.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of glycosylated hemoglobin (A1C)
Arm/Group | Sitagliptin/Metformin Fixed-Dose Combination | Pioglitazone
Number analyzed (Participants) | 253 | 246
Percent of glycosylated hemoglobin (A1C) | -1.86 [-2.00 to -1.73] | -1.39 [-1.53 to -1.26]
Statistical Analysis 1: Comparison: Sitagliptin/Metformin Fixed-Dose Combination vs Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model included a term for treatment and a covariate for the baseline A1C value; Mean Difference (Net) = -0.47, 95% CI 2-sided [-0.66 to -0.28], Standard Deviation 1.10

2. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 1
Description: Change from baseline reflects the Week 1 FPG minus the baseline FPG. At Week 1, the dose was 50/500 mg b.i.d. for Sita/Met FDC and 30 mg q.d. for pioglitazone
Time Frame: Baseline and Week 1
Population: The Full Analysis Set (FAS) included all patients who received at least one dose of double-blind study drug and had both a baseline value and ≥ 1 post-baseline value for this outcome.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin/Metformin Fixed-Dose Combination | Pioglitazone
Number analyzed (Participants) | 250 | 242
mg/dL | -40.5 [-44.1 to -36.9] | -13.0 [-16.6 to -9.3]
Statistical Analysis 1: Comparison: Sitagliptin/Metformin Fixed-Dose Combination vs Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model included a term for treatment and a covariate for the baseline FPG value; Mean Difference (Net) = -27.6, 95% CI 2-sided [-32.7 to -22.4], Standard Deviation 29.1

3. Secondary Outcome: Change From Baseline in 2-hour Post-Meal Glucose (PMG) at Week 32
Description: Change from baseline reflects the Week 32 2-hour PMG minus the baseline 2-hour PMG
Time Frame: Baseline and Week 32
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin/Metformin Fixed-Dose Combination | Pioglitazone
Number analyzed (Participants) | 192 | 198
mg/dL | -102.2 [-110.7 to -93.8] | -82.0 [-90.4 to -73.7]
Statistical Analysis 1: Comparison: Sitagliptin/Metformin Fixed-Dose Combination vs Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model included a term for treatment and a covariate for the baseline 2-hour PMG value; Mean Difference (Net) = -20.2, 95% CI 2-sided [-32.1 to -8.3], Standard Deviation 59.7

4. Secondary Outcome: Change From Baseline in FPG at Week 32
Description: Change from baseline reflects the Week 32 FPG minus the baseline FPG
Time Frame: Baseline and Week 32
Population: Full Analysis Set (FAS) included all patients who received at least one dose of double-blind study drug and had both a baseline value and ≥ 1 post-baseline value for this outcome. For FAS patients with no data at Week 32, the last non-baseline observed measurement was carried forward to Week 32.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin/Metformin Fixed-Dose Combination | Pioglitazone
Number analyzed (Participants) | 258 | 250
mg/dL | -56.0 [-60.9 to -51.0] | -44.0 [-49.1 to -39.0]
Statistical Analysis 1: Comparison: Sitagliptin/Metformin Fixed-Dose Combination vs Pioglitazone; Test type: Superiority or Other; p < 0.001, ANCOVA; ANCOVA model included a term for treatment and a covariate for the baseline FPG value; Mean Difference (Net) = -11.9, 95% CI 2-sided [-19.0 to -4.9], Standard Deviation 40.3

5. Secondary Outcome: Percent of Participants With A1C <7.0% at Week 32
Time Frame: Week 32
Population: as for outcome 1
Measure: Number; unit: Percent Participants
Arm/Group | Sitagliptin/Metformin Fixed-Dose Combination | Pioglitazone
Number analyzed (Participants) | 253 | 246
Percent Participants | 57.3 | 43.5
Statistical Analysis 1: Comparison: Sitagliptin/Metformin Fixed-Dose Combination vs Pioglitazone; Test type: Superiority or Other; p < 0.001, Regression, Logistic — Based on a test of the odds ratio = 1, comparing the odds of having A1C <7.0% at Week 32 in the Sitagliptin/Metformin 50/1000 mg b.i.d. group vs. the Pioglitazone 45 mg q.d. group; logistic regression model included a term for treatment and a covariate for the baseline A1C value; Odds Ratio (OR) = 2.0, 95% CI 2-sided [1.3 to 2.8] — This parameter estimate and 95% confidence interval correspond to the odds of having A1C <7.0% at Week 32 in the Sitagliptin/Metformin 50/1000 mg b.i.d. group vs. the Pioglitazone 45 mg q.d. group

ADVERSE EVENTS:
Time Frame: Week 0 through Week 32
Arm/Group | Sitagliptin/Metformin Fixed-Dose Combination | Pioglitazone
Serious Adverse Events (participants affected / at risk) | 11/261 | 8/256
Other Adverse Events (participants affected / at risk) | 94/261 | 68/256
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin/Metformin Fixed-Dose Combination (N=261) | Pioglitazone (N=256)
Conjunctivitis allergic (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 3 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain stem infarction (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Urine flow decreased (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sitagliptin/Metformin Fixed-Dose Combination (N=261) | Pioglitazone (N=256)
Diarrhoea (Gastrointestinal disorders) | 40 | 11
Dyspepsia (Gastrointestinal disorders) | 13 | 2
Oedema peripheral (General disorders) | 3 | 18
Nasopharyngitis (Infections and infestations) | 10 | 16
Upper respiratory tract infection (Infections and infestations) | 13 | 17
Hypoglycaemia (Metabolism and nutrition disorders) | 22 | 11
Headache (Nervous system disorders) | 20 | 7

LIMITATIONS AND CAVEATS:
Unknown to the Sponsor and the investigators, two patients in the study were randomized twice (each at two different sites). Data for these patients were deemed unreliable and excluded from all analyses (efficacy and safety).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.